CLINICAL TRIAL: NCT04422730
Title: Evolution of Body Connection and Identity Post-surgery: The Pancreas Cancer Case
Brief Title: Evolution of Body Connection After Surgery
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: COSI-PC-IPC 2019-022
Record Dates: First submitted 2019-12-02; First posted 2020-06-09 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-09

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- pancreatectomy in cancer patients
  Interventions: Behavioral: Psychological evaluation
- pancreatectomy in non-cancer patients
  Interventions: Behavioral: Psychological evaluation
- mastectomy
  Interventions: Behavioral: Psychological evaluation
- Acute leukaemia
  Interventions: Behavioral: Psychological evaluation

INTERVENTIONS:
Behavioral: Psychological evaluation — Patients will be answer to validated test about how they feel. Psychological interview is also possible depending on patients availability. The different answers will be compared between the four groups

SUMMARY:
Evaluation of psychological impact of patients after pancreatectomy because of cancer diagnosis. Patients will be evaluated with questionnaires after and before intervention. 3 control groups will be used to compare de psychological impact.

ELIGIBILITY:
Inclusion Criteria:

* Patient is older than 18 years old
* With a good understanding and practice of the French language
* And depending on the group, experimental or control, presenting:

  * pancreatic cancer expected to be treated with pancreatectomy or planned to be treated with pancreatectomy excluding cancer or breast cancer scheduled to be treated with mastectomy or acute leukaemia at a recent diagnosis (21 days).
* No patient's opposition to the information provided
* Affiliated to the social security plan or beneficiary

Exclusion Criteria:

* Other medical or psychiatric condition,
* Level of cognitive efficiency incompatible with response to questions about himself,
* A person in an emergency situation, a person under legal protection or unable to express the non opposition to their participation to research.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult people males and females
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
comparaison of Scale of Body Connection score between 4 groups | 12 months
  score from 0 to 5
comparaison of psychological interview between 4 groups | 12 months
  measured by an psychologist interpretation
comparaison of Hospital Anxiety and Dépression score between 4 groups | 12 months
  score from 0 to 21
comparaison of Test IES-R score between 4 groups | 12 months
  score from 0 to100
comparaison of quality of life score between 4 groups | 12 months
  score from 0 to 60

CONTACTS AND LOCATIONS:
Overall Officials: Thérèse AURRAN, Dr, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No